CLINICAL TRIAL: NCT02890329
Title: A Phase 1 Study of Ipilimumab in Combination With Decitabine in Relapsed or Refractory Myelodysplastic Syndrome/Acute Myeloid Leukemia
Brief Title: Ipilimumab and Decitabine in Treating Patients With Relapsed or Refractory Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01326; NCI-2016-01326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-718; 10026 (Other: Dana-Farber - Harvard Cancer Center LAO); 10026 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2025-01-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Previously Treated Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia, Myelodysplasia-Related; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine; Injections; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (decitabine, ipilimumab), post allo-HCT, Dose Level 0 (Experimental): PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Ipilimumab
- Arm A (decitabine, ipilimumab), post allo-HCT, Dose Level 1 (Experimental): PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Ipilimumab
- Arm A (decitabine, ipilimumab), post allo-HCT, Dose Level 2 (Experimental): PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Ipilimumab
- Arm B (decitabine, ipilimumab), transplant naive, Dose Level 0 (Experimental): PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Ipilimumab
- Arm B (decitabine, ipilimumab), transplant naive, Dose Level 1 (Experimental): PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Ipilimumab
- Arm B (decitabine, ipilimumab), transplant naive, Dose Level 2 (Experimental): PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Ipilimumab

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy

SUMMARY:
This phase I trial studies the side effects and best dose of ipilimumab when given together with decitabine in treating patients with myelodysplastic syndrome or acute myeloid leukemia that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ipilimumab and decitabine may work better in treating patients with relapsed or refractory myelodysplastic syndrome or acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of combination decitabine and ipilimumab for relapsed or refractory myelodysplastic syndrome (MDS) or relapsed or refractory acute myeloid leukemia (AML) in patients who are post allogeneic hematopoietic stem cell transplant (allo-HCT).

II. To determine the MTD or RP2D of combination decitabine and ipilimumab for relapsed or refractory MDS or relapsed or refractory AML in patients who are transplant naive.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the overall response rate (ORR) including complete remission (CR) and complete remission with incomplete count recovery (CRi) for AML following 2003 International Working Group (IWG) response criteria.

III. To determine the ORR including CR, partial remission, marrow CR, hematologic improvement for MDS using 2006 IWG criteria.

IV. To determine the overall survival and progression free survival at 1 year. V. To determine the duration of remission. VI. To capture the incidence and severity of acute graft-versus-host disease (GVHD) in the post allo-HCT cohort.

VII. To capture the incidence and severity of chronic graft-versus-host disease (GVHD) in the post allo-HCT cohort.

EXPLORATORY OBJECTIVES:

I. To measure the absolute lymphocyte count (ALC) prior to treatment and during treatment.

II. To evaluate the genome for evidence of clonal evolution among longitudinal samples (prior to treatment, during treatment, and at relapse if relevant) from individual patients.

III. To evaluate the histopathologic findings of immune response using immunohistochemistry.

IV. To determine the immune response in the AML tumor microenvironment by using flow cytometry and single cell mass cytometry to evaluate T cell subsets.

OUTLINE: This is a dose-escalation study of ipilimumab.

ARM A (PATIENTS POST ALLO-HCT, dose level 0):

PRIMING PHASE: Post allo-HCT patients receive decitabine intravenously (IV) over 60 minutes on days 1-5 out of 28 days.

INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM B (TRANSPLANT NAIVE PATIENTS, dose level 0):

PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.

INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM A (PATIENTS POST ALLO-HCT, dose level 1):

PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.

INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM B (TRANSPLANT NAIVE PATIENTS, dose level 1):

PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.

INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM A (PATIENTS POST ALLO-HCT, dose level 2):

PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.

INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM B (TRANSPLANT NAIVE PATIENTS, dose level 2):

PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.

INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 52 weeks (1 year).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with evidence of AML or myelodysplastic syndrome (MDS) that meet at least one of the following criteria:

  * Relapsed AML: evidence of >= 5% blasts in the bone marrow; or reappearance of blasts in the peripheral blood; or development of extramedullary disease (according to 2003 IWG criteria) who relapse after:

    * Allogeneic hematopoietic stem cell transplant, or
    * After one cycle of standard cytotoxic chemotherapy or two cycles of any hypomethylating agent-based therapy
  * Refractory AML: =< 2 prior induction regimens (example: patients who receive 7+3 followed by 5+2 would count as one induction regimen) or a minimum of two cycles of any hypomethylating agent-based therapy
  * Treatment-naive AML: must be 75 years and older with de novo or secondary AML to be considered eligible
  * Relapsed MDS: disease recurrence after CR, partial remission (PR) or hematologic improvement with bone marrow blasts >= 5% who relapse after:

    * Allogeneic hematopoietic stem cell transplant, or
    * After four cycles of any hypomethylating agent-based therapy
  * Refractory MDS: disease progression at any time after initiation of hypomethylating agent treatment or persistent bone marrow blasts >= 5% despite a minimum of four cycles of hypomethylating agent therapy
  * Untreated or previously treated therapy- related or secondary MDS
* Allowed prior allogeneic hematopoietic stem cell transplantation (allo-HCT) regardless of stem cell source; patients must be at least 3 months post allo-HCT (at time of treatment start); mismatched transplantations would be allowed
* Patients must be off systemic immunosuppressive medications > 2 weeks prior to treatment start; if patients are in systemic corticosteroids and must be on a dose of prednisone 5 mg/day or less (or equivalent), then patients must be on this reduced dose for > 1 week prior to treatment start; topical steroids are allowed
* If post allo-HCT, then patient must have baseline donor T cell chimerism of >= 20% (from peripheral blood); evaluation can be made within 4 weeks of treatment start
* No limitations on prior therapies
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x local institutional upper limit of normal (ULN)

  * If elevated total bilirubin is due Gilbert's disease or disease-related hemolysis then total bilirubin =< 3.0 x local institutional ULN
* Aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase (SGOT) =< 3.0 x local institutional ULN
* Alanine aminotransferase (ALT) or serum glutamic pyruvic transaminase (SGPT) =< 3.0 x local institutional ULN
* Serum creatinine =< 2.0 x local institutional ULN
* Negative serum pregnancy test for women who are of child bearing potential (test must be repeated if performed > 72 hours from treatment start); the effects of ipilimumab on the developing human fetus are unknown; for this reason and because immunotherapy agents as well as decitabine are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after study drug administration
* Patients with known active human immunodeficiency virus (HIV) infection; patients with chronic HIV with a CD4 > 250, undetectable viral load by polymerase chain reaction (PCR), without opportunistic infection, and on a stable regimen of highly active anti-retroviral therapy (HAART) therapy would be eligible
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 2 weeks prior to treatment start or those who have not recovered from adverse events due to agents administered more than 2 weeks prior to treatment start

  * Hydroxyurea is allowed for symptomatic leukocytosis if clinically necessary; a total white blood cell (WBC) count < 25 x 10^9/L prior to first dose of decitabine on trial is required; prior leukapheresis and/or prior or concurrent treatment with hydroxyurea to achieve this level are allowed
  * Ongoing concurrent hormonal therapy is allowed
* Participants with known central nervous system (CNS) involvement with leukemia or who are receiving intrathecal chemotherapy for active CNS leukemia

  * Those with a history of CNS involvement that has been completely treated and those who require intrathecal chemotherapy prophylaxis are eligible in the expansion cohorts
* Prior hypomethylating agent (HMA) therapy is allowed, however this study excludes patients with progression or relapse that occur while receiving HMA-based therapy within 12 weeks prior to treatment start on study; disease progression is defined as either: (1) patients with prior MDS who progress to AML (defined by the presence of >= 20% blasts in peripheral blood or bone marrow) on HMA-based therapy; OR (2) patients with AML with evidence of progressive disease according to European Leukemia Net [ELN] 2017 criteria) (e.g. > 50% increase in marrow blasts over baseline or > 50% increase in peripheral blasts to > 25 x 10^9/L (> 25,000/uL) (in absence of differentiation syndrome)

  * (Note: Patients who relapse post-transplant who received HMA treatment prior to transplant are eligible for study)
* Donor lymphocyte infusion within 8 weeks prior to treatment start if post-transplant
* For patients that are post-transplant, ineligible patients include those with a history of overall grade III or IV (severe) acute GVHD at any time even if resolved
* Patients with a history of prior treatment with anti-CTLA-4, anti-PD 1 antibody, or anti-PDL1 antibody
* Participants who are receiving any other investigational agents
* Participants with known CNS involvement with leukemia or who are receiving intrathecal chemotherapy that is either prophylactic or therapeutic; history of CNS involvement that has been completely treated (no longer receiving intrathecal chemotherapy) will be allowed
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; any other prior or ongoing condition, in the opinion of the investigator, that could adversely affect the safety of the patient or impair the assessment of study results; as patients with AML and MDS are prone to infections, if patients are actively being treated with appropriate antibiotics or antifungal therapy with clinical evidence of infection control, then they will be considered eligible for study
* Autoimmune disease: Patients who are not eligible include those with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis); patients with a history of autoimmune disease (specifically including: diabetes mellitus, vitiligo, Hashimoto's thyroiditis) who are asymptomatic, do not require immune suppression or steroids, and do not have threatened vital organ function from these conditions may be considered after discussion with the principal investigator (PI)
* No concurrent active malignancies are allowed on study for >= 2 years prior to treatment start with the exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast
* Patients with known active hepatitis B virus (HBV) infection should be excluded because of potential effects on immune function and/or drug interactions; however, if a patient has HBV history with an undetectable HBV load by polymerase chain reaction (PCR), no liver-related complications, and is on definitive HBV therapy, then he/she would be eligible for study
* Patients with known active hepatitis C virus (HCV) infection; patients with a history of HCV infection who received definitive therapy and has an undetectable viral load by PCR would be eligible
* Pregnant women are excluded from this study because ipilimumab has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ipilimumab, breastfeeding should be discontinued if the mother is treated with ipilimumab; these potential risks may also apply to decitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2026-08-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline S Garcia, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (11):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Penter L, Liu Y, Wolff JO, Yang L, Taing L, Jhaveri A, Southard J, Patel M, Cullen NM, Pfaff KL, Cieri N, Oliveira G, Kim-Schulze S, Ranasinghe S, Leonard R, Robertson T, Morgan EA, Chen HX, Song MH, Thurin M, Li S, Rodig SJ, Cibulskis C, Gabriel S, Bachireddy P, Ritz J, Streicher H, Neuberg DS, Hodi FS, Davids MS, Gnjatic S, Livak KJ, Altreuter J, Michor F, Soiffer RJ, Garcia JS, Wu CJ. Mechanisms of response and resistance to combined decitabine and ipilimumab for advanced myeloid disease. Blood. 2023 Apr 13;141(15):1817-1830. doi: 10.1182/blood.2022018246. PMID 36706355

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0: PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
- Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0: PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (3 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
- Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1: PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
- Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1: PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (5 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
- Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2: PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
- Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2: PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV (10 mg/kg) over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
Period: Cohort 1: Dose Level 0 (3 mg/kg Ipi)
Arm/Group | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2
Started | 8 | 6 | 0 | 0 | 0 | 0
Completed | 7 | 4 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progression during lead-in decitabine cycle | 1 | 1 | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 1 (5 mg/kg Ipi)
Arm/Group | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2
Started | 0 | 0 | 4 | 5 | 0 | 0
Completed | 0 | 0 | 3 | 3 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Cohort 3: Dose Level 2 (10 mg/kg Ipi)
Arm/Group | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2
Started | 0 | 0 | 0 | 0 | 15 | 16
Completed | 0 | 0 | 0 | 0 | 15 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2 | Total
Number analyzed (Participants) | 8 | 6 | 4 | 5 | 15 | 16 | 54
Age, Continuous [Median (Full Range); unit: years] | 68.5 [35 to 74] | 74.5 [59 to 82] | 64.5 [29 to 69] | 75 [50 to 81] | 66 [50 to 79] | 74.5 [34 to 85] | 71 [29 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 2 | 0 | 9 | 5 | 24
  Male | 2 | 4 | 2 | 5 | 6 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 8 | 6 | 4 | 4 | 14 | 15 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 8 | 6 | 4 | 4 | 13 | 16 | 51
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 0 | 3
ECOG Performance Status [Count of Participants; unit: Participants]
  0 (Asymptomatic and fully active) | 5 | 0 | 0 | 0 | 1 | 3 | 9
  1 (Symptomatic; fully ambulatory; restricted in physically strenuous activity) | 3 | 6 | 4 | 5 | 13 | 11 | 42
  2 (Symptomatic; ambulatory; capable of self-care greater than 50% waking hours) | 0 | 0 | 0 | 0 | 1 | 2 | 3
Histology [Count of Participants; unit: Participants]
  AML | 7 | 5 | 4 | 5 | 14 | 9 | 44
  MDS | 1 | 1 | 0 | 0 | 1 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Recommended Phase 2 Dose) of Ipilimumab in Combination With Decitabine
Description: Defined as the highest dose at which 1 or fewer of 6 patients experience a dose limiting toxicity graded by Common Terminology Criteria for Adverse Events version 5.0 criteria.
Time Frame: Monitoring for DLTs occurs continuously on treatment during the first 8 weeks of combination therapy (56 days from the start of combination) during the induction phase only.
Population: Patients who received combination ipilimumab and decitabine.
Measure: Number; unit: mg/kg
Groups:
- Arm A (Decitabine, Ipilimumab), Post Allo-HCT: PRIMING PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Post allo-HCT patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
- Arm B (Decitabine, Ipilimumab), Transplant Naive: PRIMING PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 out of 28 days.
  INDUCTION PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Transplant naive patients receive decitabine IV over 60 minutes on days 1-5 and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 4 or 8 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Ipilimumab: Given IV
Arm/Group | Arm A (Decitabine, Ipilimumab), Post Allo-HCT | Arm B (Decitabine, Ipilimumab), Transplant Naive
Number analyzed (Participants) | 25 | 23
mg/kg | 10 | 10

2. Secondary Outcome: Anti-leukemic Activity Described in Terms of Best Overall Response Rate
Description: Will be assessed by 2003 International Working Group response criteria for acute myeloid leukemia and 2006 International Working Group criteria for myelodysplastic syndrome. For acute myeloid leukemia, overall response rate includes complete remission + complete remission with incomplete count recovery; for myelodysplastic syndrome, overall response rate includes complete remission + marrow complete remission + partial remission + hematologic improvement.
Time Frame: Up to 52 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Anti-leukemic Activity Described in Terms of Progression Free Survival
Description: Will be assessed by 2003 International Working Group criteria for acute myeloid leukemia and 2006 International Working Group criteria for myelodysplastic syndrome. Time to event summaries will use the Kaplan-Meier method.
Time Frame: Time from registration to the earlier of progression or death due to any cause, assessed up to 52 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Anti-leukemic Activity Described in Terms of Overall Survival
Description: as for outcome 3
Time Frame: Time from registration to death due to any cause or censored at the date last known alive, assessed up to 52 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Acute Graft-versus-host Disease
Description: Will be separately evaluated in patients in the post-allogeneic hematopoietic stem cell transplant cohort, and compared to events with response to treatment. Graft-versus-host disease for the patients on the post-transplant arm will be estimated and reported with a 90% exact binomial confidence interval.
Time Frame: Up to 100 days
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease
Description: as for outcome 5
Time Frame: Up to 52 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Ability of Absolute Lymphocyte Count to Predict Response
Description: Absolute lymphocyte count levels will be measured prior to treatment and after cycle 2. ALC changes (from baseline to cycle 2) will be compared between responders and non-responders.
Time Frame: Up to cycle 3 day 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were continuously monitored and recorded prior to each course of therapy, from the date of registration through the date of off study, for a total of 1 lead-in and 12 combination cycles (corresponding to 52 weeks).
Description: AEs were collected by grade (using CTCAE 5.0) and treatment attribution, and max grade by toxicity type was calculated. All enrolled participants monitored/assessed for All-Cause Mortality. All participants who received at least 1 dose of ipilimumab monitored/assessed for Serious and Other (Not Including Serious) Adverse Events
Arm/Group | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2
All-Cause Mortality (participants affected / at risk) | 7/8 | 6/6 | 4/4 | 5/5 | 9/15 | 11/16
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/4 | 3/3 | 3/3 | 12/15 | 13/16
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 3/3 | 3/3 | 15/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 (N=7) | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 (N=4) | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 (N=3) | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 (N=3) | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 (N=15) | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2 (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 3 | 4 | 7
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoadrenalism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pre-septal cellulitis/Dacroadentitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Septal cellultiis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
C. diff infection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 3
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Esophageal stricutre (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
GI bleed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal Fisula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 2 | 2
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 2
Fever (General disorders) | 0 | 1 | 0 | 0 | 2 | 0
Oral GVHD (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
aGvHD (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bone infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Candidemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Central line (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
EBV reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Epstein-Barr Virus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pnemonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Strep mitis bacteria, pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Thenoorchitis epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Thenorchitis epidyditmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukemia Cutis LLE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukemia cutis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
acute on chronic subdural hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood Lactate Dehydrogenase increased (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 0 (N=7) | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 0 (N=4) | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 1 (N=3) | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 1 (N=3) | Arm A (Decitabine, Ipilimumab), Post Allo-HCT, Dose Level 2 (N=15) | Arm B (Decitabine, Ipilimumab), Transplant Naive, Dose Level 2 (N=16)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2 | 6 | 8
Bleeding from gums (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 2 | 3
Glucosuria (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphatemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Port Site Bleeding (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scraped LLL bleed (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
TSH increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transaminase elevation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 6 | 2
Tachypnea (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
heart murmur (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
mastoid cell effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Subjunctival Hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
anisocoria (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
double vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
left conjunctiva hemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
left upper eyelid stye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
stye - left upper eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
subconjunctival hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 3
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 8 | 7
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 1 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 2
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 7 | 4
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 3 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrush (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 5 | 3
pancreatic head hypodensity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
taste changes (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
AST Increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 0 | 0 | 2 | 2
Diaphoresis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 1 | 0 | 1 | 9
Edema trunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 1 | 1 | 8 | 7
Fever (General disorders) | 0 | 0 | 0 | 0 | 3 | 6
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 1 | 0 | 0 | 0 | 2 | 1
Intermittent bleeding from BMBx site (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 0 | 1 | 0 | 3 | 0
Lower Back Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Muscle cramp (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 0 | 1 | 0 | 0 | 1
Nose bleed (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 1 | 1 | 1 | 2
Rothia Mucilaginosa PICC line colonization (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transfusion reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
gallstones (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
GI GVHD (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Liver GVHD (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral GVDH (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral GVHD (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Skin GVHD (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Clostridium difficile (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
EBV Reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Epstein-Barr Virus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Thrush (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Yeast infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
neutropenic fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 1
Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Dog bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Gum bleeding (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Adrenal necrosis/Inflammatory Infiltrate (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 1 | 3 | 8
Blood bicarbonate dec. (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bicard decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 6
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
INR increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 2
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 3 | 0 | 1 | 2 | 6
Neutrophil count decreased (Investigations) | 1 | 3 | 0 | 1 | 9 | 8
Platelet count decreased (Investigations) | 2 | 2 | 0 | 3 | 6 | 7
Serum amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 1 | 0 | 0 | 1 | 5
White blood cell decreased (Investigations) | 0 | 2 | 0 | 1 | 7 | 7
increased myelofibrosis (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 8 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Glucosuria (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 5 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle Cramp (R Hand) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle Cramp (R leg) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 2
R achilles pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
muscle cramp (L leg) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
muscle cramping (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
L3 Lumbar lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 4
Dysgeusia (Nervous system disorders) | 0 | 3 | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left breast lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 4 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 3 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 5
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Erythema at PICC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0
Erythema; back (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 2 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 3 | 10
Skin GVHD (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin tear (coccyx) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
itchy skin at PICC site (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
petechial rash on BLE's (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
petechial rash on BLEs (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 3
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0 | 3 | 5
Lymphedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood Lactate Dehydrogenase increased (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 0 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT02890329/Prot_SAP_000.pdf